CLINICAL TRIAL: NCT01276236
Title: Effects of Maraviroc (MVC) on HIV-related Kaposi's Sarcoma (KS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11351; 2860798 (Other: FDA IND Exemption Reference ID)
Record Dates: First submitted 2010-12-20; First posted 2011-01-13 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Kaposi's Sarcoma
Keywords: Kaposi's Sarcoma; Maraviroc; CCR5; HIV
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Maraviroc) (Experimental): The subjects in this arm will receive Maraviroc as treatment, while continuing their current antiretroviral medication regimen.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — FDA Recommended dosing will be used in this study. Subjects on an efavirenz or etravirine-based regimen will be dosed at 600 mg orally, twice per day, for 96 weeks.
  Subjects on a ritonavir-boosted protease inhibitor based regimen (except for tipranavir/ritonavir) will be dosed at 150 mg orally, twice per day, for 96 weeks.
  Subjects that are on regimens that do not include etravirine, efavirenz, or ritonavir will be dosed at 300mg orally, twice per day, for 96 weeks. These doses are based on the recommendations from the company based on drug-drug interactions.
  Other Names: Selzentry(Celsentri outside US)

SUMMARY:
The purpose of this pilot study is to determine whether Maraviroc is effective in the treatment of Kaposi's Sarcoma (KS), when it does not remit with standard antiretroviral drug therapy.

DETAILED DESCRIPTION:
Although the advent of antiretroviral therapy (ART) may have greatly decreased the incidence of Kaposi's Sarcoma (KS) in resource rich settings, KS continues to be the most prevalent AIDS-defining malignancy in the world and carries with it significant morbidity and mortality. Indeed, in a recent epidemiological study examining cancers in Kampala, Uganda, KS was found to be second only to prostate cancer in terms of incidence rates.

There is growing evidence that C-C chemokine receptor 5 (CCR5) may be involved in the pathogenesis of KS. Kaposi's Sarcoma-associated Herpes Virus (KSHV), an agent found as necessary for KS pathogenesis, encodes viral macrophage inflammatory proteins or vMIP. vMIP-I and vMIP-II have been found to be ligands for chemokine receptors, and in particular the CCR5 receptor [5, 6], suggesting a potential role in the inflammatory process needed for KS pathogenesis. Further, vMIP-I induces Ca(2+) mobilization in monocytes expressing CCR5, suggesting an agonistic relationship between vMIP-I and the CCR5 receptor. In addition, vMIP has been found to be proangiogenic when expressed in endothelial cells, a key feature of KS tumor survival. As well, CCR5 has been found to be significantly increased in T cells populations of KS patients (from a preliminary study), and in 2 double-blind, placebo-controlled phase 3 studies in which a total of 1049 patients received the randomly assigned drug MVC, there was a trend revealing a lower incidence of KS in MVC arms vs placebo (0.36% vs 1.43%). This agonistic binding relationship between protein vMIP and CCR5, the proangiogenic activity associated with vMIP, the increased expression of CCR5 in KS, and trend towards lower incidence of KS when patients are taking MVC, suggest CCR5 may play an important role in KS pathogenesis. This involvement of CCR5 in KS pathogenesis implies that MVC may function as a potential therapeutic for KS. To date, there have been no studies examining the effect of MVC on KS.

There is a need for therapeutic development for KS. Standard of care for KS involves initiation or optimization of antiretroviral therapy. A significant proportion of KS cases do not respond to ART alone, with non-response rates ranging from 25-55%, with response times averaging 9 or more months depending on which patient series is identified. In severe or in cases of KS unresponsive to ART, standard of care involves systemic chemotherapy with liposomal doxorubicin, which is not without adverse reactions. Adverse reactions to liposomal doxorubicin include cardiac toxicity, nausea, vomiting, diarrhea, abdominal pain, fatigue, and patients may require pre-regime tests of varying costs, along with resources and time needed for intravenous infusion. Nonresponse rates for liposomal doxorubicin hover around 20%. Focal cases may be more amenable to radiation therapy or intralesional velban. However, radiation and intralesional therapies are limited to focal sites, require monitored visits and specialized care, can be given only in limited amounts, and carry various adverse effects. With these nonresponse rates, potential adverse reactions, and resources and time needed for therapeutic delivery, there are clear benefits proffered by an effective oral therapy requiring minimal monitoring, as is the case with MVC.

Maraviroc (MVC) is a member of a new class of antiretroviral compounds known as small molecule CCR5 antagonists that block R5 HIV entry into cluster of differentiation 4 (CD4) cells. Maraviroc has demonstrated selective and reversible binding to CCR5, as well as potent antiviral activity in vitro against a wide range of laboratory adapted strains of R5 HIV from Clades A, B, C, D, E, F, G, J and O. Maraviroc also retains in vitro antiviral activity against clinical isolates resistant to the existing drug classes, but has no activity against viruses that enter CD4+ cells using CXCR4. In vitro studies with approved antiretroviral medications indicate that there is no evidence of antagonism with any members of the other four classes of antiretroviral medications; nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs), non- nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors (PIs) or fusion inhibitors.

Although there is growing evidence that CCR5, a potential therapeutic target, is involved in KS pathogenesis, to date there are no studies examining the effects of a CCR5 inhibitor such as Maraviroc (MVC) on KS. As such, the aim of this study is to examine the effect of Maraviroc, a CCR5 inhibitor, on KS.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* Active biopsy confirmed KS
* Screening plasma HIV RNA < 75 copies/mL
* Patients have unremitting KS. Unremitting is defined as having active biopsy confirmed KS in spite of having had sustained HIV RNA < 75 copies/mL for 24 prior months. Isolated values that are detectable but < 500 copies will be allowed as long as the plasma HIV RNA levels before and after this time point are undetectable.
* >90% adherence to therapy within the preceding 30 days, as determined by self-report.
* Both male and female subjects are eligible. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
* Ability and willingness of subject or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Patients who are intending to modify antiretroviral therapy in the next 24 weeks for any reason.
* Serious illness requiring hospitalization or parental antibiotics within preceding 3 months.
* Concurrent treatment with immunomodulatory drugs or therapies, or exposure to any immunomodulatory drug or therapy in past 16 weeks.
* Prior exposure to CCR5 inhibitors
* Screening absolute neutrophil count <1,000 cells/mm3, platelet count <50,000 cells/mm3, hemoglobin < 8mg/dL, estimated creatinine clearance <40 mL/minute.
* Elevated transaminases greater than 2.5 times the upper limit of normal.
* Evidence of cirrhosis
* Pregnant or breastfeeding women
* Use of both Tenofovir and Didanosine in current antiretroviral therapy regimen.
* Local therapy for any KS index lesion in preceding 60 days, unless lesion has clearly progressed with enlargement since the local therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03-09 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Unemori, MD, Principal Investigator — University of California, San Francisco; San Francisco General Hospital (SFGH); Toby Maurer, MD, Principal Investigator — University of California, San Francisco; San Francisco General Hospital (SFGH)
Locations (1):
- San Francisco General Hospital, Clinical Trials Unit, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engels EA, Pfeiffer RM, Goedert JJ, Virgo P, McNeel TS, Scoppa SM, Biggar RJ; HIV/AIDS Cancer Match Study. Trends in cancer risk among people with AIDS in the United States 1980-2002. AIDS. 2006 Aug 1;20(12):1645-54. doi: 10.1097/01.aids.0000238411.75324.59. PMID 16868446
- [Background] Parkin DM, Nambooze S, Wabwire-Mangen F, Wabinga HR. Changing cancer incidence in Kampala, Uganda, 1991-2006. Int J Cancer. 2010 Mar 1;126(5):1187-95. doi: 10.1002/ijc.24838. PMID 19688826
- [Background] Gulick RM, Lalezari J, Goodrich J, Clumeck N, DeJesus E, Horban A, Nadler J, Clotet B, Karlsson A, Wohlfeiler M, Montana JB, McHale M, Sullivan J, Ridgway C, Felstead S, Dunne MW, van der Ryst E, Mayer H; MOTIVATE Study Teams. Maraviroc for previously treated patients with R5 HIV-1 infection. N Engl J Med. 2008 Oct 2;359(14):1429-41. doi: 10.1056/NEJMoa0803152. PMID 18832244
- [Background] Nakano K, Isegawa Y, Zou P, Tadagaki K, Inagi R, Yamanishi K. Kaposi's sarcoma-associated herpesvirus (KSHV)-encoded vMIP-I and vMIP-II induce signal transduction and chemotaxis in monocytic cells. Arch Virol. 2003 May;148(5):871-90. doi: 10.1007/s00705-002-0971-7. PMID 12721796
- [Background] Navenot JM, Wang ZX, Trent JO, Murray JL, Hu QX, DeLeeuw L, Moore PS, Chang Y, Peiper SC. Molecular anatomy of CCR5 engagement by physiologic and viral chemokines and HIV-1 envelope glycoproteins: differences in primary structural requirements for RANTES, MIP-1 alpha, and vMIP-II Binding. J Mol Biol. 2001 Nov 9;313(5):1181-93. doi: 10.1006/jmbi.2001.5086. PMID 11700073
- [Background] Shao W, Fernandez E, Sachpatzidis A, Wilken J, Thompson DA, Schweitzer BI, Lolis E. CCR2 and CCR5 receptor-binding properties of herpesvirus-8 vMIP-II based on sequence analysis and its solution structure. Eur J Biochem. 2001 May;268(10):2948-59. doi: 10.1046/j.1432-1327.2001.02184.x. PMID 11358512
- [Background] Nicholas J, Ruvolo VR, Burns WH, Sandford G, Wan X, Ciufo D, Hendrickson SB, Guo HG, Hayward GS, Reitz MS. Kaposi's sarcoma-associated human herpesvirus-8 encodes homologues of macrophage inflammatory protein-1 and interleukin-6. Nat Med. 1997 Mar;3(3):287-92. doi: 10.1038/nm0397-287. PMID 9055855
- [Background] Boshoff C, Endo Y, Collins PD, Takeuchi Y, Reeves JD, Schweickart VL, Siani MA, Sasaki T, Williams TJ, Gray PW, Moore PS, Chang Y, Weiss RA. Angiogenic and HIV-inhibitory functions of KSHV-encoded chemokines. Science. 1997 Oct 10;278(5336):290-4. doi: 10.1126/science.278.5336.290. PMID 9323208
- [Background] Kledal TN, Rosenkilde MM, Coulin F, Simmons G, Johnsen AH, Alouani S, Power CA, Luttichau HR, Gerstoft J, Clapham PR, Clark-Lewis I, Wells TN, Schwartz TW. A broad-spectrum chemokine antagonist encoded by Kaposi's sarcoma-associated herpesvirus. Science. 1997 Sep 12;277(5332):1656-9. doi: 10.1126/science.277.5332.1656. PMID 9287217
- [Background] Moore PS, Chang Y. Detection of herpesvirus-like DNA sequences in Kaposi's sarcoma in patients with and those without HIV infection. N Engl J Med. 1995 May 4;332(18):1181-5. doi: 10.1056/NEJM199505043321801. PMID 7700310
- [Background] Chang Y, Cesarman E, Pessin MS, Lee F, Culpepper J, Knowles DM, Moore PS. Identification of herpesvirus-like DNA sequences in AIDS-associated Kaposi's sarcoma. Science. 1994 Dec 16;266(5192):1865-9. doi: 10.1126/science.7997879.
- [Background] Cherqui S, Kingdon KM, Thorpe C, Kurian SM, Salomon DR. Lentiviral gene delivery of vMIP-II to transplanted endothelial cells and endothelial progenitors is proangiogenic in vivo. Mol Ther. 2007 Jul;15(7):1264-72. doi: 10.1038/sj.mt.6300183. Epub 2007 May 1. PMID 17505479
- [Background] Dupont C, Vasseur E, Beauchet A, Aegerter P, Berthe H, de Truchis P, Zucman D, Rouveix E, Saiag P. Long-term efficacy on Kaposi's sarcoma of highly active antiretroviral therapy in a cohort of HIV-positive patients. CISIH 92. Centre d'information et de soins de l'immunodeficience humaine. AIDS. 2000 May 26;14(8):987-93. doi: 10.1097/00002030-200005260-00010. PMID 10853980
- [Background] Nguyen HQ, Magaret AS, Kitahata MM, Van Rompaey SE, Wald A, Casper C. Persistent Kaposi sarcoma in the era of highly active antiretroviral therapy: characterizing the predictors of clinical response. AIDS. 2008 May 11;22(8):937-45. doi: 10.1097/QAD.0b013e3282ff6275. PMID 18453853
- [Background] Cooley T, Henry D, Tonda M, Sun S, O'Connell M, Rackoff W. A randomized, double-blind study of pegylated liposomal doxorubicin for the treatment of AIDS-related Kaposi's sarcoma. Oncologist. 2007 Jan;12(1):114-23. doi: 10.1634/theoncologist.12-1-114. PMID 17227906
- [Background] Cainelli F, Vallone A. Safety and efficacy of pegylated liposomal doxorubicin in HIV-associated Kaposi's sarcoma. Biologics. 2009;3:385-90. doi: 10.2147/btt.2009.3455. Epub 2009 Sep 15. PMID 19774206
- [Background] Lichterfeld M, Qurishi N, Hoffmann C, Hochdorfer B, Brockmeyer NH, Arasteh K, Mauss S, Rockstroh JK; German Clinical AIDS Working Group (KAAD). Treatment of HIV-1-associated Kaposi's sarcoma with pegylated liposomal doxorubicin and HAART simultaneously induces effective tumor remission and CD4+ T cell recovery. Infection. 2005 Jun;33(3):140-7. doi: 10.1007/s15010-005-4099-z. PMID 15940415
- [Background] Saran FH, Adamietz IA, Thilmann C, Mose S, Bottcher HD. HIV-associated cutaneous Kaposi's sarcoma--palliative local treatment by radiotherapy. Acta Oncol. 1997;36(1):55-8. doi: 10.3109/02841869709100733. PMID 9090967
- [Background] McCormick SU. Intralesional vinblastine injections for the treatment of oral Kaposi's sarcoma: report of 10 patients with 2-year follow-up. J Oral Maxillofac Surg. 1996 May;54(5):583-7; discussion 588-9. doi: 10.1016/s0278-2391(96)90637-0. PMID 8632242
- [Background] Maurer T, Ponte M, Leslie K. HIV-associated Kaposi's sarcoma with a high CD4 count and a low viral load. N Engl J Med. 2007 Sep 27;357(13):1352-3. doi: 10.1056/NEJMc070508. No abstract available. PMID 17898112

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants dosage of Maraviroc varied throughout the study depending on their non-interventional anti-viral regimen per FDA recommended dosing guidelines.
Groups:
- Treatment Arm (Maraviroc): The subjects in this arm will receive Maraviroc as treatment, while continuing their current antiretroviral medication regimen.
  Maraviroc: FDA Recommended dosing will be used in this study. Subjects on an efavirenz or etravirine-based regimen will be dosed at 600 mg orally, twice per day, for 96 weeks.
  Subjects on a ritonavir-boosted protease inhibitor based regimen (except for tipranavir/ritonavir) will be dosed at 150 mg orally, twice per day, for 96 weeks.
  Subjects that are on regimens that do not include etravirine, efavirenz, or ritonavir will be dosed at 300mg orally, twice per day, for 96 weeks. These doses are based on the recommendations from the company based on drug-drug interactions.
Period: Overall Study
Arm/Group | Treatment Arm (Maraviroc)
Started | 13
Week 36 Visit | 13
Week 56 Visit | 9
Week 76 Visit | 8
Completed | 7
Not Completed | 6
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Mean duration of Human Immunodeficiency Virus (HIV) diagnosis [Mean (Standard Deviation); unit: years] | 18.3 (2.5)
Mean duration of Kaposi's Sarcoma (KS) diagnosis [Mean (Standard Deviation); unit: years] | 7.5 (2.4)
Mean cluster of differentiation 4 (CD4) count [Mean (Standard Deviation); unit: cells in a cubic millimetre (cells/mm3)] — CD4 is a glycoprotein found on the surface of immune cells such as T helper cells, monocytes, macrophages, and dendritic cells
  cells in a cubic millimetre (cells/mm3) | 578.3 (86.3)
Number of Kaposi's Sarcoma (KS) Lesions at Baseline [Count of Participants; unit: Participants]
  >50 lesions | 4
  <=50 lesions | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in Kaposi's Sarcoma (KS) Total Surface Area
Description: To assess improvements in disease, up to five bi-dimensionally measurable cutaneous KS lesions were selected as marker lesions. The collective surface area of the marker lesions was evaluated over the course of the study for either an increase or decrease in the total surface area of lesions using the modified AIDS Clinical Trials Group (ACTG) Oncology Committee Staging Criteria.
Time Frame: Up to 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 13
Participants | 11

2. Primary Outcome: Percent Change in KS Total Surface Area
Description: Up to five bi-dimensionally measurable cutaneous KS lesions were selected as marker lesions and the the collective surface area of the marker lesions was evaluated over the course of the study. The percent decrease or increase in the total surface area of lesions was calculated from comparing measurements at baseline and through week 96, or at the last assessment if participant withdrew from the study prior to week 96.
Time Frame: Up to 96 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 13
percentage change | -28.1 (7.9)

3. Primary Outcome: Change in Edema Grade
Description: The presence and extent of lower extremity edema was assessed and graded on a scale from 0 to 2 in patients with a higher grade indicating a greater level of edema using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS Adverse Events (AE) Grading Table), Version 1.0. Edema grade was recorded at baseline was compared with edema grades recorded at week 96, or at last assessment if participant withdrew from study prior to week 96 and an change in grade was calculated to examine whether or not a decrease in overall grade was observed. A negative value would indicate an overall decrease in the grade of lower extremity edema, and positive value would indicate an overall increase in lower extremity edema.
Time Frame: Up to 96 weeks
Population: Only seven patients total had measurable edema at any time during the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 7
scores on a scale | -0.7 (0.3)

4. Secondary Outcome: Change in Kaposi's Sarcoma-associated Herpesvirus (KSHV) Viral Load
Description: Blood and saliva samples will be obtained from the subjects throughout the study at different points to assess if there are any changes in KSHV viral load.
Time Frame: Up to 96 weeks
Population: Data was not collected for this endpoint
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 0

5. Secondary Outcome: Percent Change in CCR5 Levels on CD4+ T-Cells
Description: Maraviroc works by binding to the C-C chemokine receptor 5 (CCR5) on T-cells and thereby blocking viral entry into CD4+ T-cells. Peripheral blood mononuclear cells (PBMC) were obtained from blood draws at each visit and T-cell immunophenotyping was performed from the baseline visit and final follow-up visit to determine the percent change in CCR5 levels on CD4+ T-Cells
Time Frame: Up to 96 weeks
Population: Only 5 participants had greater than 80% cell viability in peripheral blood mononuclear cell (PBMC) specimens required for flow cytometry at baseline and final follow-up.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 5
percentage change | 22.8 (5.9)

6. Secondary Outcome: Percent Change in CCR5 Levels on CD8+ T-cells
Description: Maraviroc works by binding to the C-C chemokine receptor 5 (CCR5) on T-cells and thereby blocking viral entry into CD8+ T-cells. Peripheral blood mononuclear cells (PBMC) were obtained from blood draws at each visit and T-cell immunophenotyping was performed from the baseline visit and final follow-up visit to determine the percent change in CCR5 levels on CD8+ T-Cells
Time Frame: Up to 96 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 5
percentage change | 21.6 (3.5)

7. Secondary Outcome: Percent Change in CD69 Expression in a Subset of Double Negative DR-CD38 Positive (DR-CD38+) T-cells
Description: Peripheral blood mononuclear cells (PBMC) were obtained from blood draws at each visit and T-cell immunophenotyping was performed from the baseline visit and final follow-up visit to determine the percent change in CD69 expression in a subset of double negative DR-CD38 positive (DR-CD38+) T-cells
Time Frame: Up to 96 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 5
percentage change | 89.7 (48.2)

8. Secondary Outcome: Percent Change in CD69 Expression in a Subset of Double Negative DR-CD38 Negative (DR-CD38-) T-cells
Description: Peripheral blood mononuclear cells (PBMC) were obtained from blood draws at each visit and T-cell immunophenotyping was performed from the baseline visit and final follow-up visit to determine the percent change in CD69 expression in a subset of double negative DR-CD38- T-cells
Time Frame: Up to 96 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment Arm (Maraviroc)
Number analyzed (Participants) | 5
percentage change | 50.5 (35.9)

ADVERSE EVENTS:
Time Frame: Up to 96 weeks
Description: No grade 3 or higher adverse events were reported during study. Participants dosage of Maraviroc varied throughout the study depending on their non-interventional anti-viral regimen per FDA recommended dosing guidelines. Dosing was not held or limited based on low-grade adverse events therefore adverse event data was aggregated across all dosages.
Arm/Group | Treatment Arm (Maraviroc)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 12/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (Maraviroc) (N=13)
Fatigue (General disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 5 participants had greater than 80% cell viability in peripheral blood mononuclear cell (PBMC) specimens required for flow cytometry at baseline and final follow-up. In the remaining eight patients, either the baseline or final follow-up or both specimens had lower than 80% cell viability and were therefore excluded from immunophenotyping analyses. The small sample sizes reduced the statistical power of the reported results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes